CLINICAL TRIAL: NCT03336437
Title: The Impact of Local Estrogen on the Urogenital Microbiome in Genitourinary Syndrome of Menopause (GSM)
Brief Title: Estrogen and the Urogenital Microbiome in GSM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jennifer Lillemon, House Officer, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OHSU IRB# 17056
Record Dates: First submitted 2017-11-02; First posted 2017-11-08 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-09

CONDITIONS: Menopause
Keywords: Menopause; Vaginal dryness; Vaginal atrophy; Postmenopause; Estrogen; Urinary microbiome; Estradiol vaginal ring; Genitourinary Syndrome of Menopause; Vaginal microbiome

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estrogen Vaginal Ring (Active Comparator): At the time of initial study visit, a estrogen vaginal ring (Estring) will be placed. Participants will retain this ring for 12 weeks.
  Interventions: Drug: Estradiol vaginal ring
- Inactive Vaginal Placebo Ring (Placebo Comparator): At the time of initial study visit, a placebo vaginal ring will be placed. Participants will retain this ring for 12 weeks.
  Interventions: Other: Placebo vaginal ring

INTERVENTIONS:
Drug: Estradiol vaginal ring — Estradiol 2mg vaginal ring
  Arms: Estrogen Vaginal Ring
Other: Placebo vaginal ring — Silicone vaginal ring without any active estradiol
  Arms: Inactive Vaginal Placebo Ring

SUMMARY:
This is a study of how local estrogen treatment affects the microbiome of the vagina and bladder in postmenopausal women experiencing symptoms as part of "Genitourinary Syndrome of Menopause." The goal is to understand more about the underlying microbial changes occurring in menopause and whether these are reversible with estrogen.

DETAILED DESCRIPTION:
Women who have undergone menopause almost ubiquitously experience pelvic complaints at some point in the postmenopausal period. This is most commonly vaginal dryness and discomfort during sexual intercourse. From previous studies, we know that as estrogen levels decrease in menopause, changes occur in the local urogenital tract that include thinning of the vaginal epithelium, an increase in pH and an alteration of the composition of the local bacterial community, including a decrease in the typically predominant species of bacteria lactobacilli. In conjunction with declining estrogen levels, a subset of postmenopausal women experience bothersome lower urinary tract symptoms such as burning with urination, urinary urgency, incontinence and recurrent urinary tract infections. These symptoms are commonly underreported, under-treated, and have been associated with reduced quality of life and decreased productivity in menopause. "Genitourinary Syndrome of Menopause" (GSM) is a term adapted to be more inclusive of these lower urinary tract symptoms in an effort to reduce delays in evaluation and treatment. It remains controversial whether these symptoms relate directly to estrogen deprivation or are part of the "natural" aging process. Mainstay therapy includes vaginal lubricants and local estrogen therapy. Though treatment with local estrogen improves both vaginal dryness as well as urinary symptoms, the mechanism is not well understood.

Additionally, there is a subset of women who do not respond to estrogen treatment or have contraindications to estrogen use. Recent research efforts have been exploring the potential role that the microbiome may play in female pelvic discomfort and dysfunction. Unlike the vagina, the bladder has historically been considered to be a sterile environment, with the presence of bacteria implying infection. However, recent research has helped to elucidate that, similar to the skin, vagina and gastrointestinal tract, a resident microbial community or "microbiome" exists within the female bladder. Disturbances in the urinary microbial community have been correlated with conditions such as painful bladder syndrome, overactive bladder and urge urinary incontinence. These conditions have considerable symptom overlap with those seen in postmenopausal women who are experiencing GSM and may be considered to be on the same continuum.

Though microbiome research over the last decade has accelerated our understanding of the role that organisms play in health and disease, the urinary microbiome remains poorly defined. Data from ongoing research suggests that the urinary microbiome of pre- and postmenopausal women differ, which would suggest that hormone status may play a role in maintaining the microbial milieu. This research has helped us to better understand how the urinary microbiome varies under normal conditions. In order to better understand the role that estrogen plays in maintaining the bladder and vaginal flora, this study aims to characterize the effect of local estrogen on the urinary and vaginal microbiomes (together termed the "urogenital microbiome") in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female
* Generally healthy

Exclusion Criteria:

* Known allergy or contraindications to the intervention
* Use of hormone therapy in the last 3 months
* Current tamoxifen use
* Currently using vaginal pessary
* History of breast cancer or BRCA mutation
* History of uterine, ovarian or cervical cancer
* History of deep vein thrombosis or pulmonary embolism
* History of stroke or myocardial infarction
* Known thrombophilic disorder (Protein S deficiency, Protein C deficiency, antithrombin deficiency)
* Known liver disease
* Use of systemic or vaginal antibiotics in the last 2 months
* Urinary tract or vaginal infection in the last 2 months

Ages: 40 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Urinary Microbiome: change in the relative abundance of urinary lactobacillus between baseline and 12 weeks post intervention | Baseline to 12 weeks post-intervention
  Investigators will collect catheterized urine samples from participants at time of enrollment in the study and again after 12 weeks of their assigned vaginal ring intervention. Bacteria will be extracted from the urine and the resident microbial community will be characterized by amplifying the bacterial 16S ribosomal RNA gene via PCR. The de-identified samples containing amplified 16S DNA will be sequenced using Illumina MiSeq. The genetic sequences will be processed to generate a table of bacterial identity and relative quantity. Statistical tests designed for microbiome data will be used in order to determine differences between the relative amount of lactobacillus (via the lactobacillus ratio) before and after the intervention.

SECONDARY OUTCOMES:
Change in prevalence of GSM symptoms | Baseline to 12 weeks post-intervention
  Validated symptom questionnaires will be collected at baseline and again after 12 weeks of assigned intervention to assess common symptoms associated with Genitourinary Syndrome of Menopause (GSM), such as vaginal dryness, painful intercourse and urinary urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lillemon, Principal Investigator — Oregon Health and Science University
Locations (1):
- Women's Health Research Unit at Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lillemon JN, Karstens L, Nardos R, Garg B, Boniface ER, Gregory WT. The Impact of Local Estrogen on the Urogenital Microbiome in Genitourinary Syndrome of Menopause: A Randomized-Controlled Trial. Female Pelvic Med Reconstr Surg. 2022 Jun 1;28(6):e157-e162. doi: 10.1097/SPV.0000000000001170. Epub 2022 Apr 15. PMID 35420551